CLINICAL TRIAL: NCT00255281
Title: A Double-Blind, Randomised, Placebo-Controlled, Parallel-Group, Multicentre, Phase II Study to Assess the Efficacy of AZD7009 (AR H065522XX) Given Intravenously (Infusion for 15 or 30 Minutes) to Patients for Conversion of Atrial Fibrillation
Brief Title: Efficacy and Safety of AZD7009 in the Treatment of Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1461C00006
Record Dates: First submitted 2005-11-17; First posted 2005-11-18 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — AZD 7009

INTERVENTIONS:
Drug: AZD7009, no generic name available

SUMMARY:
The current study is designed to assess the efficacy and safety of iv AZD7009 in conversion from AF

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for cardioversion of Atrial Fibrillation. Effective oral anticoagulation according to local routines or a TEE without any finding of intracardial thrombus or signs of thrombogenecity

Exclusion Criteria:

* Clinically significant sinus and/or AV node dysfunction. Serum or plasma potassium <3.8 mmol/L or >5.0 mmol/L. QTc(Bazett) >450 ms. Any QRS duration >150 ms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2005-09; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The proportion of patients that have converted from AF within 90 minutes from start of infusion.

SECONDARY OUTCOMES:
The time to conversion of AF from start of the infusion.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AZD7009 Midical Science Director, MD, Study Director — AstraZeneca
Locations (32):
- Denmark (4):
  - Research Site, Esbjerg
  - Research Site, Hellerup
  - Research Site, Hvidovre
  - Research Site, Svendborg
- Finland (2):
  - Research Site, Helsinki
  - Research Site, Oulu
- Germany (6):
  - Research Site, Aachen
  - Research Site, Bad Berka
  - Research Site, Brandenburg
  - Research Site, Hamburg
  - Research Site, Magdeburg
  - Research Site, Münster
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Kecskemét
  - Research Site, Szentes
  - Research Site, Székesfehérvár
- Netherlands (3):
  - Research Site, Groningen
  - Research Site, Maastricht
  - Research Site, Stadskanaal
- Norway (4):
  - Research Site, Oslo
  - Research Site, Rud
  - Research Site, Tromsø
  - Research Site, Trondheim
- Poland (5):
  - Research Site, Bytom
  - Research Site, Opole
  - Research Site, Ruda Śląska
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Sweden (3):
  - Research Site, Linköping
  - Research Site, Örebro
  - Research Site, Stockholm